CLINICAL TRIAL: NCT02750540
Title: DREAM-01: Optimization of a Tenofovir Enema for HIV Prevention
Brief Title: Optimization of a Tenofovir Enema for HIV Prevention
Acronym: DREAM-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of California, Los Angeles (Other); University of Pittsburgh (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00097186; DAIDS ES 12067 (Other: NIAID/ DAIDS); 5U19AI113127 (NIH)
Record Dates: First submitted 2016-04-11; First posted 2016-04-25 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: HIV Prevention
Keywords: Tenofovir enema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Product A dose (Active Comparator): Product A will contain tenofovir (TFV) 220 mg in 125 mL iso-osmolar solution: Participants will have a single dose administered in clinic or a research unit, followed by various specimen collections over 8 days, according to individual sampling schedule assigned to each participant; specimens will be collected on Day 1, 2, 4, and 8.
  Interventions: Drug: Tenofovir enema
- Product B dose (Active Comparator): Product B will contain tenofovir (TFV) *660 mg in 125 mL iso-osmolar solution: Participants will have a single dose administered in clinic or a research unit, followed by various specimen collections over 8 days, according to individual sampling schedule assigned to each participant; specimens will be collected on Day 1, 2, 4, and 8.
  Interventions: Drug: Tenofovir enema
- Product C dose (Active Comparator): Product C will contain tenofovir (TFV) *660 mg in 125 mL hypo-osmolar solution at half the osmolarity of iso-osmolar solution: Participants will have a single dose administered in clinic or a research unit, followed by various specimen collections over 8 days, according to individual sampling schedule assigned to each participant; specimens will be collected on Day 1, 2, 4, and 8.
  Interventions: Drug: Tenofovir enema
- Take-home normal saline (NS) enema (Placebo Comparator): The normal saline (NS) solution will be provided following administration of Product A which is iso-osmolar. The volume of NS enema (120 mL) was selected to approximately match that of Product A (125 mL)
  Interventions: Other: Saline enema
- Take-home half normal saline (½ NS) enema (Placebo Comparator): The ½ normal saline (½ NS) solution will be provided following administration of Product C which is hypo-osmolar. The volume of the ½ NS enema (120 mL) was selected to approximately match that of Product C (125 mL)
  Interventions: Other: Saline enema

INTERVENTIONS:
Drug: Tenofovir enema
  Arms: Product A dose; Product B dose; Product C dose
Other: Saline enema
  Arms: Take-home half normal saline (½ NS) enema; Take-home normal saline (NS) enema

SUMMARY:
DREAM-01 is an early phase 1, open label, dose-escalation and variable osmolarity study to compare the safety, pharmacokinetics (PK), pharmacodynamics (PD), and acceptability of 3 formulations of a tenofovir (TFV) enema. The goal of the study is to identify the dose and osmolarity of a TFV enema for human immunodeficiency virus (HIV) pre-exposure prophylaxis (PrEP) which achieves the desired colonic mucosal mononuclear cells (MMC) tenofovir diphosphate (TFV-DP) target concentrations that have previously been shown to confer protection from HIV acquisition in men who have sex with men (MSM).

DETAILED DESCRIPTION:
DREAM-01 is an early phase 1, open label, dose-escalation and variable osmolarity study to compare the safety, pharmacokinetics (PK), pharmacodynamics (PD), and acceptability of 3 formulations of a tenofovir (TFV) enema. The goal of the study is to identify the dose and osmolarity of a TFV enema for human immunodeficiency virus (HIV) pre-exposure prophylaxis (PrEP) which achieves the desired colonic mucosal mononuclear cells (MMC) tenofovir diphosphate (TFV-DP) target concentrations that have previously been shown to confer protection from HIV acquisition in men who have sex with men (MSM).

Each participant will undergo screening to evaluate eligibility. Baseline visit will assess safety, PD, and behavioral readout baselines. Three products described below (Product A, B, and C) are dosed sequentially as a dose-escalation within each subject. Safety, PK, PD, and behavioral readouts are assessed at specified times for one week after each dose, followed by a variable washout period before the next escalation dose. Johns Hopkins University (JHU) participants only will have SPECT/CT imaging to assess distribution and permeability of radiolabeled product. After two of the study product doses (Product A and Product C) and their respective sampling periods, a normal saline (NS) solution and ½ normal saline (½ NS) solution will be taken at home in the context of receptive anal intercourse.

Study Duration: Participant accrual will take approximately 9 months and each participant will be on study for approximately 4-5 months. Total study duration is about 1 year.

Study Products: Three study products administered sequentially and estimated to approximate TFV 1% gel (Product A), 3 times the concentration and dose of Product A (Product B), and 2 times concentration and dose of Product B (Product C) as defined below. At JHU only, the study product will also be radiolabeled with Technetium-99m-DTPA (99mTc-DTPA) for SPECT/CT imaging. Take-home enemas consisting of normal saline (NS) or ½ normal saline (½ NS) will be self-administered at home.

* Product A: Enema formulation of TFV 1.76 mg/mL (220 mg in 125 mL) in iso-osmolar solution
* Product B: Enema formulation of TFV 5.28 mg/mL (*660 mg in 125 mL) in iso-osmolar solution
* Product C: Rectal specific Enema formulation of TFV 5.28 mg/mL (*660 mg in 125 mL) in hypo-osmolar solution
* Take-home enema to follow Product A: 120 mL of normal saline (NS) solution
* Take-home enema to follow Product C: ½ normal saline (½ NS)

  * Note: the planned 660 mg TFV dose in Product B and C may be adjusted lower or higher based on Product A results in order to more closely achieve target concentrations - this is indicated by *660 mg, which will be used throughout the protocol to indicate the planned, but potentially modified Product B (or C as the case may be) dose.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older at screening
2. Willing and able to communicate in English
3. Willing and able to provide written informed consent to take part in the study
4. Willing and able to provide adequate locator information
5. Understand and agree to local Sexually Transmitted Infection (STI) reporting requirements
6. Biologically male
7. HIV-1 uninfected at screening as documented by Combo Ag/Ab HIV-1/HIV-2 immunoassay (refer to Appendix II for confirmatory testing algorithm)
8. Available to return for all study visits, barring unforeseen circumstances
9. Per participant report at screening, a history of consensual Receptive Anal Intercourse (RAI) at least five times in lifetime and at least once in the prior 3 months (Required to ensure that participants are sufficiently sexually active to complete take-home enema study requirements)
10. Per participant report at screening, experience with receiving or self-administering an enema or douche in the past year.
11. Willing to abstain from insertion of anything (drug/medication, penis, object, sex toy, or enema including take-home enema) into the anorectum for 72 hours before and after each research unit study product exposure and 7 days after each flexible sigmoidoscopy with biopsy collection.
12. Willing to refrain from aspirin and NSAID use for one week before and after each study biopsy visit
13. Willing and able to use condoms provided by the study for all Receptive Anal Intercourse (RAI) for the duration of participation
14. Agrees not to participate in other research studies involving drugs and/ or medical devices for the duration of the study

Exclusion Criteria:

1. History of chronic Hepatitis B infection, as documented by positive HBsAg at screening
2. ≥ Grade 2 laboratory abnormality at baseline as defined by The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0 dated November 2014
3. Significant colorectal symptom(s) as determined by medical history or by participant self-report (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, history of inflammatory bowel disease, presence of symptomatic external hemorrhoids, and presence of any painful anorectal conditions that would be tender to manipulation)
4. At screening or within the past 2 months: participant-reported symptoms and/or clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include Chlamydia (CT), gonorrhea (GC), syphilis, active Herpes Simplex Virus (HSV) lesions, chancroid, genital sores or ulcers, and, if clinically indicated, genital warts. Note that HSV seropositivity with no active genital lesions is not an exclusion criterion, since treatment is not required.
5. History of an underlying cardiac arrhythmia or renal disease (including creatinine clearance <50 mL/min using Cockcroft-Gault equation)
6. History of severe or recent cardiac or pulmonary event
7. History of aortic aneurysm
8. History of significant gastrointestinal bleeding
9. Current use of warfarin or heparin or other anticoagulant medications associated with increased risk for bleeding following mucosal biopsy (e.g., daily high dose aspirin [>81 mg], NSAIDs, or Pradaxa®)
10. Use of systemic or anorectal immunomodulatory medications within 4 weeks of enrollment or planned use at any time during study participation
11. Use of pre-exposure (PrEP) and post-exposure (PEP) prophylaxis for HIV exposure within 3 weeks of enrollment or planned use within 3 weeks prior to any study visit with PK sampling.
12. Per participant report, use of any rectally administered products containing N-9 (including condoms) or investigational products within 4 weeks of enrollment, or planned use of either at any time during study participation
13. Known allergic reaction to TFV or other components of the test articles
14. Current known HIV-infected partners
15. History of recurrent urticaria
16. For JHU only: Participants whose whole body (Effective Dose Equivalent or EDE) radiation exposure, per the investigator's records and/or participant report, exceeds 5000 Millirem (mRem)/year
17. Symptoms suggestive of acute HIV seroconversion at screening and enrollment
18. Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events Grade 2 or higher, using Division of AIDS Adverse Events Grading Tables | A total number of adverse events will be assessed through study completion, time period of up to 9 months
  Adverse events occurring between dosing and day 7 for each of 3 doses during the study (each will be assessed as a unique dose related event period lasting 7 days) will be assessed according to the following scale: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-Threatening
Area under the curve of tenofovir concentration matrix at 1 hr post dose | 1 hr post dose
  TFV-DP concentration will be measured at 1 hr post dose in order to assess target concentrations in colonic mucosal mononuclear cells (MMC) for each study product
Area under the curve of tenofovir concentration matrix at 3 hr post dose | 3 hr post dose
  TFV-DP concentration will be measured at 3 hr post dose in order to assess target concentrations in colonic mucosal mononuclear cells (MMC) for each study product
Area under the curve of tenofovir concentration matrix at 6 hr post dose | 6 hr post dose
  TFV-DP concentration will be measured at 6 hr post dose in order to assess target concentrations in colonic mucosal mononuclear cells (MMC) for each study product
Area under the curve of tenofovir concentration matrix at 12 hr post dose | 12 hr post dose
  TFV-DP concentration will be measured at 12 hr post dose in order to assess target concentrations in colonic mucosal mononuclear cells (MMC) for each study product
Area under the curve of tenofovir concentration matrix at 24 hr post dose | 24 hr post dose
  TFV-DP concentration will be measured at 24 hr post dose in order to assess target concentrations in colonic mucosal mononuclear cells (MMC) for each study product
Area under the curve of tenofovir concentration matrix at 72 hr post dose | 72 hr post dose
  TFV-DP concentration will be measured at 72 hr post dose in order to assess target concentrations in colonic mucosal mononuclear cells (MMC) for each study product
Area under the curve of tenofovir concentration matrix at 168 hr post dose | 168 hr post dose
  TFV-DP concentration will be measured at 168 hr post dose in order to assess target concentrations in colonic mucosal mononuclear cells (MMC) for each study product
Proportion of subjects who consider the tenofovir study products acceptable for use as assessed by a behavioral questionnaire | After each TFV enema product (at 1 to 6 hours post dose)
  For each product, descriptive statistics of overall product acceptability will be generated (i.e., mean and standard deviation for continuous variables and proportion of subjects who consider the products acceptable -- with score 3 or greater). In addition, a futility test will be conducted for each product to screen out non-acceptable product(s) and identify the product(s) with potential for being acceptable to users in a future study. The acceptability of each product is defined as a mean score of 3 on 4-point continuous acceptability measure (1=completely unacceptable; 2=somewhat unacceptable; 3=somewhat acceptable; 4=highly acceptable) that is defined in this study as the minimal clinically meaningful threshold for product acceptability.
Proportion of subjects who consider using the saline enemas at home acceptable as assessed by a behavioral questionnaire | Within 30 days after completing the low dose TFV enema use and high dose TFV enema use in clinic
  Descriptive statistics of overall product acceptability will be generated (i.e., mean and standard deviation for continuous variables and proportion of subjects who consider the products acceptable -- with score 3 or greater). In addition, a futility test will be conducted for each product to screen out non-acceptable product(s) and identify the product(s) with potential for being acceptable to users in a future study. The acceptability of each product is defined as a mean score of 3 on 4-point continuous acceptability measure (1=completely unacceptable; 2=somewhat unacceptable; 3=somewhat acceptable; 4=highly acceptable) that is defined in this study as the minimal clinically meaningful threshold for product acceptability.
Proportion of subjects who consider all enema study products acceptable for use as assessed by a behavioral questionnaire | At the end of each subject's study participation, after all 3 products have been administered in clinic and at home, which is up to 1 month after the last product is administered at home. The total period of study depends on interim data analysis.
  Descriptive statistics of overall product acceptability will be generated (i.e., mean and standard deviation for continuous variables and proportion of subjects who consider the products acceptable -- with score 3 or greater). In addition, a futility test will be conducted for each product to screen out non-acceptable product(s) and identify the product(s) with potential for being acceptable to users in a future study. The acceptability of each product is defined as a mean score of 3 on 4-point continuous acceptability measure (1=completely unacceptable; 2=somewhat unacceptable; 3=somewhat acceptable; 4=highly acceptable) that is defined in this study as the minimal clinically meaningful threshold for product acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Ethel D Weld, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Center for Prevention Research, University of California Los Angeles, Los Angeles, California
  - The Johns Hopkins University, Baltimore, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giguere R, Balan IC, Lentz C, Dolezal C, Carballo-Dieguez A, Fuchs EJ, Anton P, McGowan I, Ho K, Weld E, Hendrix CW. Acceptability of a rectal microbicide douche for HIV prevention: a mixed-methods analysis of a first-in-human formulation pilot study. Sex Transm Infect. 2025 Jan 29;101(1):49-54. doi: 10.1136/sextrans-2024-056209. PMID 39237135
- [Derived] Weld ED, McGowan I, Anton P, Fuchs EJ, Ho K, Carballo-Dieguez A, Rohan LC, Giguere R, Brand R, Edick S, Bakshi RP, Parsons T, Manohar M, Seigel A, Engstrom J, Elliott J, Jacobson C, Bagia C, Wang L, Al-Khouja A, Hartman DJ, Bumpus NN, Spiegel HML, Marzinke MA, Hendrix CW. Tenofovir Douche as HIV Preexposure Prophylaxis for Receptive Anal Intercourse: Safety, Acceptability, Pharmacokinetics, and Pharmacodynamics (DREAM 01). J Infect Dis. 2024 Apr 12;229(4):1131-1140. doi: 10.1093/infdis/jiad535. PMID 38019657